CLINICAL TRIAL: NCT05784103
Title: Measurement of Oxygen Saturation in Healthy Human Volunteers Before, During, and After Hyperemic Events Using Multi-Modal Techniques: Spatial Frequency Domain Imaging, Transcutaneous Oxygen Measurement, Pulse Oximeter, and Apple Watch
Brief Title: Comparison of Tissue Oxygenation Measurement Using Multimodal Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Surya Gnyawali, Asst. Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13895
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Results first posted 2023-11-24 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Oxygen Saturation
Keywords: SFDI, oxygenation, healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Multi-Modal Measurement of Oxygen Saturation (Other): During a single study visit, participants will have oxygen saturation measured with a number of oximetry devices including Spatial Frequency Domain Imaging (SFDI), Transcutaneous oxygen monitoring (TCOM), an Apple Watch Oxygen Sensor, and a Pulse Oximeter. Each device will be used to measure oxygen saturation of the thumb and index fingers at rest, during occlusion of blood flow to the arm (using an inflated blood pressure cuff applied to the arm), and during the hyperemic post-occlusion period. Completion of all planned interventions may take up to 2 hours on the study visit day.
  Interventions: Device: Clarifi Modulum; Device: Perimed PeriFlux 5000; Device: Apple Watch Oxygen Sensor; Device: Innovo iP 900AP

INTERVENTIONS:
Device: Clarifi Modulum — During consenting period, the Modulim equipment will be calibrated and setup ready for scanning. Subject's volar aspect of the thumb along with the palm surface will be ready to target the optical camera head. Actual scanning takes less than 60 seconds. The images will be processed offline. During processing 3-5 different regions of interest will be taken to measure the oxygen parameters such as tissue oxygen saturation, oxy-hemoglobin, deoxy-hemoglobin, superficial hemoglobin, and sub-surface hemoglobin.
  Other Names: Spatial Frequency Domain Imaging (SFDI)
Device: Perimed PeriFlux 5000 — Transcutaneous oxygen monitoring (TCOM or TcpO2) is a noninvasive, clinically-approved method to obtain skin oxygen levels. The method is quantitative, and measures oxygen delivery to the skin from underlying tissue. Before positioning the electrode, an adhesive fixation ring will be placed on the dry skin on the volar aspect of the thumb and an electrolyte as a contact liquid will be filled half and the probe is aligned into it by rotating clock-wise to fasten it. Recording will be started and waited for the oxygen level to stabilize and a fixed value will be recorded. The probe will be heated to about 45oC. Although this device has other options, only the measurement of O2 will be performed using this device.
  Other Names: Transcutaneous oxygen monitoring (TCOM)
Device: Apple Watch Oxygen Sensor — The apple watch is equipped with green, red, and infrared LEDs that shine light onto the blood vessels in the wrist, with photodiodes measuring the amount of light reflected back. Apple's algorithms use this information to calculate the color of the blood, which is an indication of how much oxygen is in the blood. Bright red blood is well oxygenated, while darker blood has less oxygen. This can measure blood oxygen levels between 70 and 100 percent. Most healthy people have blood oxygen levels that range from 95 to 100 percent. The apple watch sensor will be positioned on the user's preferred wrist.
Device: Innovo iP 900AP — The pulse oximeter enables transcutaneous monitoring of the oxygen saturation of hemoglobin in arterial blood. In this study, volar aspect of thumb and index finder of the subject will be used to measure blood oxygen saturation.
  Other Names: Pulse Oximeter

SUMMARY:
Pulse oximeters are common medical devices used to measure blood oxygen saturation (SpO2). These devices are either stand-alone or integrated into physiologic monitoring systems, using 2 wavelengths of light to determine SpO2. With recent advances in technology, Spatial Frequency Domain Imaging (SFDI) uses a range of light wavelengths from red to near-infrared (NIR), and smartphones such as Apple Watch, and transcutaneous oximetry TCOM now have pulse oximetry capabilities. Since it is possible that most patients could utilize this technology, we sought to assess the accuracy, reliability, and usability of these oximeters and compare outcomes. In this study, a cohort of 20 healthy volunteers above the age of 18 including males and females of different skin colors will be assessed at the same site and data will be compared. We aim to provide a set of data that will support the clinical and scientific community and identify more than one reliable skin oxygen measurement modality.

DETAILED DESCRIPTION:
The subjects will go through a questionnaire session about their medical history by a designated study team member. The questionnaire data will be placed in RedCap using a subject ID that cannot be linked back to the subject. Then the subject will consent and be enrolled. Then the non-invasive data-collecting procedure will start on the following equipment.

Spatial Frequency Domain Imaging (SFDI): During the consenting period, the Modulim equipment will be calibrated and set up ready for scanning. The subject's volar aspect of the thumb along with the palm surface will be ready to target the optical camera head. Actual scanning takes less than 60 seconds. The images will be processed offline. During processing 3-5 different regions of interest (ROI) will be taken to measure the oxygen parameters such as tissue oxygen saturation (StO2), oxy-hemoglobin (HbO2), deoxy-hemoglobin (HbR), superficial hemoglobin (HbT1, sub-surface hemoglobin (HbT2). The model used is a Clarifi Modulim Transcutaneous oxygen monitoring (TCOM): Transcutaneous oxygen monitoring (TCOM or TcpO2) is a noninvasive, clinically-approved method to obtain skin oxygen levels. The method is quantitative and measures oxygen delivery to the skin from underlying tissue. Before positioning the electrode, an adhesive fixation ring will be placed on the dry skin on the volar aspect of the thumb and an electrolyte as a contact liquid will be filled in half and the probe is aligned into it by rotating clockwise to fasten it. The recording will be started and waited for the oxygen level to stabilize and a fixed value will be recorded. The model used is a Perimed PeriFlux 5000. The probe will be heated to about 45 degrees C. Although this device has other options, only the measurement of O2 will be performed using this device.

Apple Watch Oxygen Sensor: Smartwatch blood oxygen sensors also measure blood oxygen levels in the tissue. Apple Watch Series 6 introduced this new feature for monitoring blood oxygen levels using light-emitting diodes (LEDs) at the back of apple watches. A low blood oxygen level can be indicative of a serious health issue that needs immediate attention. The apple watch is equipped with green, red, and infrared LEDs that shine light onto the blood vessels in the wrist, with photodiodes measuring the amount of light reflected back. Apple's algorithms use this information to calculate the color of the blood, which is an indication of how much oxygen is in the blood. Bright red blood is well-oxygenated, while darker blood has less oxygen. This can measure blood oxygen levels between 70 and 100 percent. Most healthy people have blood oxygen levels that range from 95 to 100 percent. The apple watch sensor will be positioned on the user's preferred wrist.

Pulse Oximeter for Oxygen Monitoring: The pulse oximeter enables transcutaneous monitoring of the oxygen saturation of hemoglobin in arterial blood (StO2). Pulse oximetry is so widely prevalent in medical care that it is often regarded as a fifth vital sign[3]. It is important to understand how the technology functions as well as its limitations. To recognize the settings in which pulse oximeter readings of oxygen saturation (SpO2), an understanding of two basic principles of pulse oximetry is required: (i) how oxyhemoglobin (HbO2) is distinguished from deoxyhemoglobin (HbR) and (ii) how the SpO2 is calculated only from the arterial compartment of blood. Pulse oximetry is based on the principle that HbO2 and HbR differentially absorb red and near-infrared (IR) light. It is fortuitous that HbO2 and HbR have significant differences in absorption at red and near-IR light because these two wavelengths penetrate tissues well whereas blue, green, yellow, and far-IR light are significantly absorbed by non-vascular tissues and water [3]. HbO2 absorbs greater amounts of IR light and lower amounts of red light than does HbR; this is consistent with experience - well-oxygenated blood with its higher concentrations of HbO2 appears bright red to the eye because it scatters more red light than does HbR. On the other hand, HHR absorbs more red light and appears less red. Exploiting this difference in light absorption properties between HbO2 and HbR, pulse oximeters emit two wavelengths of light, red at 660 nm and near-IR at 940 nm from a pair of small light-emitting diodes located in one arm of the finger probe. The light that is transmitted through the finger is then detected by a photodiode on the opposite arm of the probe. In this study, the volar aspect of the thumb and index finger of the subject will be used to measure SpO2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Able to understand and complete the Informed Consent
* Both males and females
* Age between 18-65 years
* All ethnic backgrounds

Exclusion Criteria:

* Patients or limited health conditions
* Smoking tobacco product
* Prisoners
* Cannot consent for themselves

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Surya C. Gnyawali, PhD, Principal Investigator — University of Pittsburgh and Indiana University, School of Medicine
Locations (2):
- United States (2):
  - Indiana University, School of Medicine, Indianapolis, Indiana
  - Surya C. Gnyawali, University of Pittsburgh, UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Through Publication

REFERENCES:
- [Result] Jones MD, Taylor JL, Barry BK. Occlusion of blood flow attenuates exercise-induced hypoalgesia in the occluded limb of healthy adults. J Appl Physiol (1985). 2017 May 1;122(5):1284-1291. doi: 10.1152/japplphysiol.01004.2016. Epub 2017 Feb 9. PMID 28183823
- [Derived] El Masry M, Li R, Balasubramani GK, Roy S, Sen CK, Gnyawali SC. Comparative assessment of healthy tissue oxygenation using near-infrared imaging, transcutaneous oxygen measurement, and plethysmography. Sci Rep. 2025 Aug 19;15(1):30424. doi: 10.1038/s41598-025-15767-2. PMID 40830190

RESULTS

PARTICIPANT FLOW:
Groups:
- Multi-modal Measurement of Tissue Oxygenation: SFDI: StO2= tissue oxygen saturation HbO2=oxy hemoglobin HbR= deoxyhemoglobin HbT1= superficial perfusion hemoglobin HbT2= deep perfusion hemoglobin TCOM=trans-cutaneous oxygen measurement SFDI=spatial frequency domain imaging
Period: Overall Study
Arm/Group | Multi-modal Measurement of Tissue Oxygenation
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All 20 participants were taken for baseline. Before the occlusion was considered baseline and after the occlusion was compared before occlusion as baseline for each patient.
Groups:
- Multi-Modal Measurement of Tissue Oxygenation on Healthy Volunteers: In a single study visit, oxygen saturation was measured on participants with SFDI, TCOM, Apple Watch Oxygen Sensor, and a Pulse Oximeter. The thumb and index fingers are at rest, during the occlusion, and during the hyperemic post-occlusion period. Completion of all planned interventions may take up to 2 hours on the study visit day.
  Modulum: Equipment will be calibrated and set up ready for scanning. volar aspect of the thumb surface imaged. parameters: tissue oxygen saturation, oxy-hemoglobin, deoxy-hemoglobin, superficial hemoglobin, and sub-surface hemoglobin.
  PeriFlux 5000: tcpO2 is a noninvasive, clinically-approved method to obtain skin oxygen levels. The probe is placed on dry skin on the volar aspect of the thumb. A recording will be started and waited for the oxygen level to stabilize and a fixed value will be recorded.
  Apple Watch Oxygen Sensor: The Apple watch wrist's Bright red blood is well-oxygenated, while darker blood has less oxygen. Can measure blood oxygen levels between 70 and 100 percent. Healthy people have blood oxygen levels that range from 95 to 100 percent.
  Oximeter: The pulse oximeter enables monitoring of the oxyhemoglobin in arterial blood. volar aspect index finder of the subject was used to measure blood oxygen saturation.
Arm/Group | Multi-Modal Measurement of Tissue Oxygenation on Healthy Volunteers
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (6.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Device-wise Comparison of Tissue Oxygenation Measurement
Description: 4 devices used to measures the tissue oxygen saturation on healthy human volunteers
Time Frame: Visit 1, up to 2 hours in duration
Population: The Apple watch and the Pulse Oximeters are the devices designed to measure blood oxygenation based on the blood pulses occurring in the blood vessels when there is actual flow. At the time of occlusion there is no blood vessels pulsating, so the data were measured zero.
Measure: Mean (Standard Deviation); unit: percentage of oxygen
Groups:
- SFDI: During a single study visit, participants will have oxygen saturation measured with Spatial Frequency Domain Imaging (SFDI). measure oxygen saturation of the thumb and index fingers at rest, during occlusion of blood flow to the arm (using an inflated blood pressure cuff applied to the arm), and during the hyperemic post-occlusion period. Completion of all planned interventions may take up to 2 hours on the study visit day.
- TCOM: During a single study visit, participants will have oxygen saturation measured with TCOM. measure oxygen partial pressure of the thumb and index fingers at rest, during occlusion of blood flow to the arm (using an inflated blood pressure cuff applied to the arm), and during the hyperemic post-occlusion period. Completion of all planned interventions may take up to 2 hours on the study visit day.
- Apple Watch: During a single study visit, participants will have oxygen saturation measured with the Apple Watch application. measure oxygenation of the thumb and index fingers at rest, during occlusion of blood flow to the arm (using an inflated blood pressure cuff applied to the arm), and during the hyperemic post-occlusion period. Completion of all planned interventions may take up to 2 hours on the study visit day.
- Pulse Oximeter: During a single study visit, participants will have oxygen saturation measured with Pulse Oximeter. measure oxygenation of the thumb and index fingers at rest, during occlusion of blood flow to the arm (using an inflated blood pressure cuff applied to the arm), and during the hyperemic post-occlusion period. Completion of all planned interventions may take up to 2 hours on the study visit day.
Arm/Group | SFDI | TCOM | Apple Watch | Pulse Oximeter
Number analyzed (Participants) | 20 | 20 | 20 | 20
percentage of oxygen
  baseline | 62.7 (18.11) | 91.2 (11.98) | 97.58 (1.14) | 97.95 (1.05)
  during occlusion | 44.8 (16.03) | 67.95 (14.97) | 0 (0) | 0 (0)
  reactive hyperamia | 71.1 (17.41) | 87.21 (9.09) | 97.88 (1.16) | 99.24 (1.09)
  Recovery | 65.8 (17.94) | 79.9 (10.70) | 97.50 (1.12) | 97.56 (1.04)

2. Primary Outcome: Male vs Female Comparison of Tissue Oxygenation Measurement
Description: Goal is to see if there is a variation in the gender biased. The criteria for the male vs female comparison were considered to find better or worse outcomes.
Time Frame: 1 visit, 2hrs
Population: The Apple watch and the Pulse Oximeters are the devices designed to measure blood oxygenation based on the blood pulses occurring in the blood vessels when there is actual flow. At the time of occlusion there is no blood flow, the vessels are not pulsating, so the data were measured zero.
Measure: Mean (Standard Deviation); unit: percentage of Oxygen
Groups:
- SFDI Measurement of Oxygen Saturation: Modulum: Modulim calibrated and set up ready for scanning. volar aspect of the thumb surface to target the optical camera head. oxygen parameters tissue oxygen, oxy-hemoglobin, deoxy-hemoglobin, superficial hemoglobin, and sub-surface hemoglobin.
- PeriFlux 5000 for Transcutaneous Oxygen Partial Pressure: PeriFlux 5000: tcpO2 is a noninvasive, clinically-approved method to obtain skin oxygen levels. The method is quantitative and measures oxygen delivery to the skin from underlying tissue. The probe was heated to about 45 deg C. Although this device has other options, only the measurement of O2 will be performed using this device.
- Apple Watch Oxygen Sensor for Arterial Oxygenation: Apple Watch Oxygen Sensor: Apple watch is equipped with green, red, and infrared LEDs that shine light onto the blood vessels in the wrist. This can measure blood oxygen levels between 70 and 100 percent. Most healthy people have blood oxygen levels that range from 95 to 100 percent. Apple watch sensor will be positioned on the user's preferred wrist.
- A Pulse Oximeter for Arterial Oxygenation: Innovo iP 900AP: The pulse oximeter enables transcutaneous monitoring of the oxygen saturation of hemoglobin in arterial blood. In this study, volar aspect of thumb and index finder of the subject will be used to measure blood oxygen saturation.
Arm/Group | SFDI Measurement of Oxygen Saturation | PeriFlux 5000 for Transcutaneous Oxygen Partial Pressure | Apple Watch Oxygen Sensor for Arterial Oxygenation | A Pulse Oximeter for Arterial Oxygenation
Number analyzed (Participants) | 20 | 20 | 20 | 20
percentage of Oxygen
  Male: number analyzed (Participants) | 13 | 13 | 13 | 13
  Male | 61.40 (21.75) | 94.15 (10.67) | 97.43 (1.00) | 97.87 (0.91)
  Female: number analyzed (Participants) | 7 | 7 | 7 | 7
  Female | 65.48 (6.48) | 85.61 (14.54) | 97.85 (0.96) | 98.09 (0.62)

3. Primary Outcome: Skin Type Based Comparison of Tissue Oxygenation
Description: Fitzpatrick chart-based skin categorization of the skin type. The criteria for the Fitzpatrick Skin Type grades IV, II & III were matched with Fitzpatric table and grades were considered to find better or worse outcomes.
  Please Note: The skin type analysis was performed irrespective to the devices. Only skin types were considered. So, there is no need of adding arms/groups other than the (1) Skin type IV and (2) the skin type II& III.
Time Frame: 1 visit, 2hrs duration
Population: Type II: Fitzpatrick grades were according to the following criteria:- Fair skin, blue eyes; burns easily, tans poorly.
  Type III: Fitzpatrick grades were according to the following criteria:- Darker white skin; tans after initial burn.
  Type IV: Fitzpatrick grades were according to the following criteria:- Light brown skin; burns minimally, tans easily.
  This was used to grade from the Fitzpatrick skin type scale questionnaire.
Measure: Mean (Standard Deviation); unit: percentage of oxygen
Groups:
- Fitzpatrick Skin Type IV Based Analysis: a plastic surgeon assessed the skin and based on Fitzpatrick chart; the skin-types were identified. Completion of interventions took up to 20 minutes on the study visit day. Higher scores were placed in group IV.
- Fitzpatrick Skin Type II & III: a plastic surgeon assessed the skin and based on Fitzpatrick chart; the skin-types were identified. Completion of interventions took up to 20 minutes on the study visit day. lower scores were placed in group II and III.
Arm/Group | Fitzpatrick Skin Type IV Based Analysis | Fitzpatrick Skin Type II & III
Number analyzed (Participants) | 7 | 13
percentage of oxygen | 21.62 (3.09) | 24.64 (2.66)

ADVERSE EVENTS:
Time Frame: up to 1 week
Description: They are healthy volunteers
Arm/Group | SFDI Measurement of Oxygen Saturation | PeriFlux 5000 for Transcutaneous Oxygen Partial Pressure | Apple Watch Oxygen Sensor for Arterial Oxygenation | A Pulse Oximeter for Arterial Oxygenation
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
The study includes a small cohort of 20 volunteers. Aim was to include dark skin volunteers but that was not successful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/03/NCT05784103/Prot_003.pdf
  • Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/03/NCT05784103/SAP_004.pdf
  • Informed Consent Form (2022-02-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT05784103/ICF_006.pdf